CLINICAL TRIAL: NCT04742400
Title: A Phase 2 Clinical Trial of Tolebrutinib, a Brain-penetrant Bruton's Tyrosine Kinase Inhibitor, for the Modulation of Chronically Inflamed White Matter Lesions in Multiple Sclerosis
Brief Title: Tolebrutinib, a Brain-penetrant Bruton's Tyrosine Kinase Inhibitor, for the Modulation of Chronically Inflamed White Matter Lesions in Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210010; 21-N-0010
Record Dates: First submitted 2021-02-05; First posted 2021-02-08 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-05-08

CONDITIONS: Multiple Sclerosis
Keywords: MS; BTK Inhibitor
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tolebrutinib (Cohort A) (Experimental): Tolebrutinib 60 mg/day for 48 weeks, Tolebrutinib 120 mg/day for 96 weeks
  Interventions: Drug: tolebrutinib 60mg; Drug: tolebrutinib 120mg
- Tolebrutinib (cohort B) (Experimental): Tolebrutinib 120 mg daily
  Interventions: Drug: tolebrutinib 120mg
- tolebrutinib (initial cohort) (Experimental): Tolebrutinib 60 mg daily
  Interventions: Drug: tolebrutinib 60mg

INTERVENTIONS:
Drug: tolebrutinib 60mg — 60 mg orally
  Arms: Tolebrutinib (Cohort A); tolebrutinib (initial cohort)
Drug: tolebrutinib 120mg — 120 mg orally
  Arms: Tolebrutinib (Cohort A); Tolebrutinib (cohort B)

SUMMARY:
Background:

Some multiple sclerosis (MS) lesions stay inflamed for very long periods of time. This type of inflammation is not affected by any MS medications. These lesions can lead to slow worsening of MS symptoms. Researchers want to see if a new drug can help.

Objective:

To see if tolebrutinib can help clear inflammation in MS brain lesions.

Eligibility:

Adults ages 18 and older with MS who are on an anti-CD20 therapy.

Design:

Participants will be screened under protocol #89-N-0045.

Participants will have a medical history. They will have physical and neurological exams. They will have blood and urine tests. The progression of their MS will be assessed.

Participants will have MRIs of the brain. The MRI scanner is shaped like a cylinder. It uses a magnetic field and radio waves to take pictures of the body. During the MRIs, participants will lie on a table that slides in and out of the scanner. Soft padding or a coil will be placed around their head.

Participants may have electrocardiograms to measure the heart s electrical activity.

Participants may have lumbar punctures ( spinal taps ). A small needle will be inserted into the spinal canal in the lower back. Fluid will be collected.

Some participants will take tolebrutinib pills by mouth once a day for at least 96 weeks. They will stop their anti-CD20 therapy. They will have at least 10 study visits.

Some participants will not take tolebrutinib. They will stay on their anti-CD20 therapy. They will have 5 study visits.

Participation will last at least 96 weeks.

DETAILED DESCRIPTION:
Study Description:

The primary goal of this protocol is to test whether 48 weeks of treatment with tolebrutinib, an investigational, orally available, brain-penetrant, Bruton's tyrosine kinase (BTK) inhibitor, affects an imaging marker (the paramagnetic rim) associated with chronically inflamed white matter lesions in multiple sclerosis (MS). In this rater-blinded but otherwise open- label study, 16 adults with MS who are on stable disease-modifying treatment with anti-CD20 antibody therapy and are within 6 months of their most recent dose, have at least one paramagnetic rim lesion on 7-tesla magnetic resonance imaging (MRI), and have developed no new white matter lesions or clinical relapses for at least 6 months, will initiate treatment with tolebrutinib and agree to forego further anti- CD20 or other disease-modifying therapy for the duration of the trial.

An initial 7 enrolled study participants started tolebrutinib at 60 mg/day (Initial Cohort). Of the Initial Cohort, participants (n=3), who had initiated tolebrutinib 60 mg will remain at 60 mg and not be escalated to 120 mg/day. The remaining participants (n=4) consented to Cohort A, who had initiated tolebrutinib 60 mg and previously escalated to 120 mg/day will remain at that dose.

Radiological, clinical, and biological outcomes are measured at 24, 48, 72, 96, and 144 (Cohort A) weeks, with additional interspersed visits for safety monitoring. Participants may subsequently continue treatment until tolebrutinib is marketed or commercial development halted. A comparison group of 10 participants who meet enrollment criteria but choose to stay on anti-CD20 therapy will also be enrolled. The primary outcome measure is disappearance of one or more paramagnetic rims from white matter lesions identified at baseline. Secondary outcomes include safety and tolerability and additional radiological outcomes. Exploratory clinical, radiological, and laboratory investigations are planned to study the mechanism of action of tolebrutinib and for biomarker development, and to compare the tolebrutinib and anti-CD20 cohorts.

Objectives:

Primary Objective: To evaluate the effects of 48 weeks of tolebrutinib 60 mg/day treatment on the paramagnetic rim of chronically inflamed white matter lesions, as seen on 7-tesla MRI.

Secondary Objectives: (1) To assess safety and tolerability of 48 weeks of treatment with tolebrutinib 60 mg and 96 weeks of treatment with tolebrutinib 120 mg (Cohort A) all following anti-CD20 antibody therapy. (2) To assess the possible repair of chronically inflamed white matter lesions in which inflammation at the lesion edge has been modulated by tolebrutinib.

Endpoints:

Primary Endpoint: Per-patient proportion of lesions in which the paramagnetic rim has disappeared at the end of 48 weeks of tolebrutinib 60 mg.

Secondary Endpoints: (1) Adverse event tables. (2) Changes in T1 relaxation time within paramagnetic rim lesions at the end of 96 weeks of tolebrutinib 120 mg, relative to non-rim lesions. (3) Changes in size of paramagnetic rim lesions at the end of 96 weeks of tolebrutinib 120 mg, relative to non-rim lesions.

Study Population:

Up to 10 adults with multiple sclerosis, targeting at least 7 participants who complete 48 weeks of therapy with tolebrutinib 60 mg in Cohort A. Up to 10 adults with multiple sclerosis who meet inclusion criteria but choose to stay on anti-CD20 therapy.

Phase 2:

Description of Study Intervention:

Oral tolebrutinib 60 mg per day for 48 weeks (Initial Cohort), and a subgroup of patients already escalated to 120 mg (Cohort A), with optional long-term extension and follow-up.

Study Duration:

5 years

Participant Duration:

144 weeks (Cohort A) for primary and secondary outcomes, with optional long-term extension and follow-up.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Tolebrutinib Cohorts Inclusion Criteria

1. Able to provide informed consent
2. Willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged greater than or equal to 18
4. Diagnosed with multiple sclerosis according to the 2017 revision of the McDonald diagnostic criteria, with no new lesion formation by comparison of baseline MRI scan with a historical MRI scan at least 6 months prior
5. On anti-CD20 antibody treatment for at least 6 months, with the most recent dose at most 6 months prior to enrollment.
6. Willing to forego further anti-CD20 antibody treatment for the duration of the study
7. Fully vaccinated against SARS-CoV-2 by Day 0. At the time of this writing, Fully vaccinated is defined as:

   * Two weeks out from the second dose of a two-dose vaccine series (Moderna, Pfizer-BioNTech); or
   * Two weeks out from a single-dose vaccine (Johnson & Johnson/Janssen)
   * Note: Should guidelines change, we will amend these inclusion criteria accordingly
8. Has a prior 7-tesla MRI scan, no more than 1 year prior to enrollment, demonstrating at least one white matter lesion with a paramagnetic rim
9. For females of reproductive potential: agrees to use highly effective contraception for at least 1 month prior to dosing and to use such a method during study participation and for an additional 12 weeks after the end of tolebrutinib administration
10. For males of reproductive potential: agrees to use condoms or other methods to ensure effective contraception with partner; agrees not to donate sperm from the inclusion up to 12 weeks after the last dose
11. QuantiFERON-TB Gold negative; skin testing (e.g., tuberculin skin test) will be allowed if blood testing is not available or the blood test result is indeterminate
12. Agrees to adhere to Lifestyle Considerations throughout study duration
13. Agrees not to participate in any other interventional study while participating in this protocol

Control Cohort Inclusion Criteria:

1. Able to provide informed consent
2. Willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged greater than or equal to 18
4. Diagnosed with multiple sclerosis according to the 2017 revision of the McDonald diagnostic criteria, with no new lesion formation by comparison of baseline MRI scan with a historical MRI scan at least 6 months prior
5. On anti-CD20 antibody treatment for at least 6 months, with the most recent dose at most 6 months prior to enrollment. (Participants in this cohort should remain on their baseline anti-CD20 treatment at least through week 48.)
6. Has a prior 7-tesla MRI scan, no more than 1 year prior to enrollment, demonstrating at least one white matter lesion with a paramagnetic rim
7. For females of reproductive potential: agrees to use highly effective contraception during study participation
8. Agrees not to participate in any other interventional study while participating in this protocol

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

Tolebrutinib Cohorts Exclusion Criteria

1. Pregnancy or lactation
2. MS relapse in the 6 months prior to dosing
3. Febrile illness within 4 weeks prior to dosing, or persistent chronic or active infection requiring treatment with systemic antibiotics, antivirals, or antifungals.
4. Treatment with another investigational drug or other investigational intervention within 3 months prior to baseline
5. Contraindications for 7-tesla MRI
6. Presence of screening laboratory or ECG values outside normal limits that are considered in the PI or MAI s judgment to be clinically significant, including but not limited to:

   1. Presence of liver injury defined as underlying hepatobiliary disease or screening alanine aminotransferase (ALT) more than 1.5 times the upper limit of normal (ULN)
   2. At screening, positive for hepatitis B surface antigen and/or hepatitis B core antibody and/or positive for hepatitis C antibody
   3. Any of the following:

      * Bleeding disorder or known platelet dysfunction at any time prior to the first screening visit
      * Platelet count less than 150,000/microL at the screening visit
   4. Lymphocyte count less than 1000 cells/dL at the screening visit
7. Is HIV-positive
8. Has received any live (attenuated) vaccine (including but not limited to varicella zoster, oral polio, and nasal influenza) within 2 months before dosing
9. Has received any of the following medications/treatments within the specified time frame before baseline assessment:

   * Medication: Systemic corticosteroids, adrenocorticotropic hormone (other than used for premedication); Exclusionary if used/used within required wash-out period: 1 month prior to baseline MRI scan
   * Medication: Dimethyl fumarate; Exclusionary if used/used within required wash-out period: 6 months prior to dosing
   * Medication: Intravenous immunoglobulin, fingolimod, natalizumab; Exclusionary if used/used within required wash-out period: 6 months prior to dosing
   * Medication: Teriflunomide; Exclusionary if used/used within required wash-out period: 2 years prior to dosing or 1 month prior to dosing

   if participant undergoes an accelerated elimination procedure and has documented teriflunomide plasma level below 0.02 mg/L

   before dosing
   * Medication: Mildly to moderately immunosuppressive/chemotherapeutic medications such azathioprine and methotrexate; Exclusionary if used/used within required wash-out period: 6 months prior to dosing
   * Medication: Highly immunosuppressive/chemotherapeutic medications: mitoxantrone up to 120 mg/m2 body surface area, cyclophosphamide, cladribine; Exclusionary if used/used within required wash-out period: 2 years prior to dosing
   * Medication: Alemtuzumab; Exclusionary if used/used within required wash-out period: 4 years prior to dosing
   * Medication: Lymphoid irradiation, bone marrow transplantation, mitoxantrone (with evidence of cardiotoxicity following treatment, or cumulative lifetime dose >120 mg/m2), other strongly immunosuppressive treatments with very long-lasting effects; Exclusionary if used/used within required wash-out period: Any time
   * Medication: Any BTK inhibitor; Exclusionary if used/used within required wash-out period: Any time
10. Is receiving potent and moderate inducers and inhibitors of cytochrome P450 3A (CYP3A) or potent inhibitors of CYP2C8 hepatic enzymes.
11. Is receiving anticoagulant/antiplatelet therapies, including:

    1. Acetylsalicylic acid (aspirin); half-life elimination: Parent drug: Plasma concentration: 15 to 20 minutes; Salicylates (dose dependent): 3 hours at lower doses (300 to 600 mg), 5 to 6 hours (after 1 g), 10 hours with higher doses
    2. Antiplatelet drugs (eg, clopidogrel); half-life: 6 hours
    3. Warfarin (vitamin K antagonist); half-life: 20-60 hours
    4. Heparin, including low molecular weight heparin (antithrombin agents); half-life: 60-90 minutes
    5. Dabigatran (direct thrombin inhibitor); half-life:12-17 hours
    6. Apixaban (IV half-life: approximately 5 hours, oral half-life: approximately 12 hours), edoxaban (half-life: 10-14 hours), rivaroxaban (half-life: 5-9 or 11-13 hours in younger or elderly individuals, respectively) (direct factor Xa inhibitors)

    Note: All above drugs need to be stopped at least 5 half-lives before study drug administration except for aspirin, which needs to be stopped at least 8 days before.
12. Has a history or presence of significant other concomitant illness that, according to the PI or MAI s judgment, would adversely affect participation in this study; examples include but are not limited to clinically significant cardiovascular, renal, hepatic, or metabolic

    disease.
    * Acute liver disease, cirrhosis, chronic liver disease (unless considered stable for >6 months)
    * Has untreated hepatitis C
    * Has chronic hepatitis B unless stable on oral suppression and/or followed by a local hepatologist to monitor for reactivation
    * Has active alcohol use disorder
    * Has an alcohol intake greater than 2 drink per day for men, and greater than 1 drink per day for women (1 drink = approximately 14 grams of alcohol = 350 ml beer = 140 mL wine = 40 mL of spirits)
    * Has aspartate transaminase (AST) or alanine transaminase (ALT) levels greater than 1.5x ULN
    * Has a total bilirubin level greater than 1.5x ULN unless due to Gilbert s or non-liver related disorder
    * Has an alkaline phosphatase level greater than 2x ULN unless caused by non-liver related disorder or explained by a stable chronic liver disorder
    * At baseline, elevated transferrin saturation (>50% in males and >40% in females) and/or with elevated ferritin levels >500 microgram/L.
13. Unwilling to allow coded samples to be processed offsite
14. Unwilling to have coded samples and/or data saved or used in other studies.

Control Cohort Exclusion Criteria:

1. Pregnancy or lactation
2. MS relapse in the 6 months prior to baseline
3. Treatment with another investigational drug or other investigational intervention within 3 months prior to baseline
4. Contraindications for 7-tesla MRI
5. Has received any of the following medications/treatments within the specified time frame before baseline assessment:

   * Medication: Systemic corticosteroids, adrenocorticotropic hormone (other than used for premedication); Exclusionary if used/used within required wash-out period: 1 month prior to baseline MRI scan
   * Medication: Dimethyl fumarate; Exclusionary if used/used within required wash-out period: 6 months prior to dosing
   * Medication: Intravenous immunoglobulin, fingolimod, natalizumab; Exclusionary if used/used within required wash-out period: 6 months prior to dosing
   * Medication: Teriflunomide; Exclusionary if used/used within required wash-out period: 2 years prior to dosing or 1 month prior to dosing if participant undergoes an accelerated elimination procedure and has documented teriflunomide plasma level below 0.02 mg/L before dosing
   * Medication: Mildly to moderately immunosuppressive/chemotherapeutic medications such azathioprine and methotrexate; Exclusionary if used/used within required wash-out period: 6 months prior to dosing
   * Medication: Highly immunosuppressive/chemotherapeutic medications: mitoxantrone up to 120 mg/m2 body surface area, cyclophosphamide, cladribine; Exclusionary if used/used within required wash-out period: 2 years prior to dosing
   * Medication: Alemtuzumab; Exclusionary if used/used within required wash-out period: 4 years prior to dosing
   * Medication: Lymphoid irradiation, bone marrow transplantation, mitoxantrone (with evidence of cardiotoxicity following treatment, or cumulative lifetime dose >120 mg/m2), other strongly immunosuppressive treatments with very long-lasting effects; Exclusionary if used/used within required wash-out period: Any time
   * Medication: Any BTK inhibitor; Exclusionary if used/used within required wash-out period: Any time
6. Has a history or presence of significant other concomitant illness that, according to the PI or MAI s judgment, would adversely affect participation in this study; examples include but are not limited to clinically significant cardiovascular, renal, hepatic, or metabolic

   disease.
7. Unwilling to allow coded samples to be processed offsite
8. Unwilling to have coded samples and/or data saved or used in other studies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD that results in a publication
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: IPD will be shared under tech transfer agreements.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2021-N-0010.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with MS were recruited between April 1, 2021 and November 30, 2023. Participants were referred by both internal and external providers, and were self-referred.
Groups:
- Tolebrutinib Cohort: Participants on Tolebrutinib 60 mg/day for 48 weeks.
- Anti-CD20 Cohort: Participants on baseline Anti-CD20 continuing at least through week 48.
Period: Overall Study
Arm/Group | Tolebrutinib Cohort | Anti-CD20 Cohort
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolebrutinib Cohort | Anti-CD20 Cohort | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.7 (7.8) | 42 (6.11) | 45.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 6 | 3 | 9
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
Paramagnetic Rim Lesions [Median (Full Range); unit: Number of Paramagnetic Rim Lesions] | 9 [6 to 46] | 4.5 [2 to 7] | 8 [2 to 46]

OUTCOME MEASURES:

1. Primary Outcome: Disappearance of Paramagnetic Rim Lesions at 48 Weeks of 60 mg of Tolebrutinib.
Description: Paramagnetic rims indicate the presence of inflammation and ongoing demyelination and axonal transection at the lesion edge. The lesions under study were present for at least 6 months. The results represent the number of participants in whom at least the paramagnetic rim has disappeared in at least 1 lesion at the end of 48 weeks of tolebrutinib 60 mg.
Time Frame: 48 weeks
Measure: Number; unit: Participants
Arm/Group | Tolebrutinib Cohort | Anti-CD20 Cohort
Number analyzed (Participants) | 7 | 5
Participants | 0 | 0

2. Secondary Outcome: Safety and Tolerability of Tolebrutinib.
Description: To assess safety and tolerability of 96 weeks of tolebrutinib 60 mg (initial cohort), or 48 weeks of treatment with tolebrutinib 60 mg and 96 weeks off treatment with tolebrutinib 120 mg (Cohort A), all following anti-CD20antibody.
Time Frame: each patient visit
Reporting Status: Not Posted

3. Secondary Outcome: Repair of Chronically Inflamed White Matter Lesions
Description: To assess the possible repair of chronically inflamed white matter lesions in which inflammation at the lesion edge has been modulated by tolebrutinib. A reduction of the T1 relaxation time would be compatible with lesion repair. A reduction in lesion size could indicate lesion repair.
Time Frame: baseline vs. 96 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Tolebrutinib Cohort | Anti-CD20 Cohort
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/5
Other Adverse Events (participants affected / at risk) | 7/7 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolebrutinib Cohort (N=7) | Anti-CD20 Cohort (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tolebrutinib Cohort (N=7) | Anti-CD20 Cohort (N=5)
Asymptomatic conduction disorder (Cardiac disorders) | 2 (2) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Tinnitus
Presbyopia (Eye disorders) | 1 (1) | 0 (0) — Presbyopia
Subconjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0) — Subconjunctival hemorrhage
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Diarrhea
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) — Nausea
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) — Oral hemorrhage
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Stomach pain
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bruising (worsening) (General disorders) | 1 (1) | 0 (0)
Facial pain (left side) (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Peripheral edema (General disorders) | 1 (1) | 0 (0)
Acute upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2)
Bruising and/or other injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Mechanical fall (skiing) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Right 2nd digit and right foot laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Elevated white blood cell count in cerebrospinal fluid (Investigations) | 0 (0) | 1 (1)
Hypokalemia, grade 1 (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscus tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bilateral lower extremity paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leak (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Increased tingling in right upper extremity (Nervous system disorders) | 0 (0) | 1 (1)
Left leg heaviness (Nervous system disorders) | 1 (1) | 0 (0)
Leg weakness (Nervous system disorders) | 1 (1) | 0 (0)
New lesion (Nervous system disorders) | 0 (0) | 1 (1)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Weakness (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Vivid dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Renal and urinary disorders other: hesitancy (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin lesion/insect bite (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-03): https://cdn.clinicaltrials.gov/large-docs/00/NCT04742400/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT04742400/ICF_001.pdf